CLINICAL TRIAL: NCT02016391
Title: Effects of Dexmedetomidine on Periprocedural Pain During Radiofrequency Ablation of Liver and Kidney Tumours
Brief Title: Effects of Dexmedetomidine During Radiofrequency Ablation of Abdominal Tumours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Egidijus Semenas, Consultant in anaesthesia and intensive care, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF-01; 2013/409 (Other: Uppsala Regional Ethics Committee)
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Cancer of Kidney and Renal Pelvis; Cancer of Liver
MeSH Terms: conditions — Kidney Neoplasms; Liver Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.4 µg/kg/hr infusion during RF procedure

SUMMARY:
The purpose of he study is to evaluate effects of dexmedetomidine on pain during radiofrequency ablation of liver and kidney tumours.

DETAILED DESCRIPTION:
Although radiofrequency ablation (RF) is accepted as the best therapeutic choice for patients with early stage hepatocellular carcinoma when liver transplantation or surgical resection are not suitable options, it is still performed only in a few hospitals and experience is so far limited (Goldberg & Ahmed, 2002; Shiina et al., 2005). In addition, RF ablation is emerging as a viable alternative to surgery for inoperable patients with limited hepatic metastatic disease, especially from colorectal cancer. Although radiofrequency ablation has been accepted as a safe and effective treatment for liver and kidney tumours, there are few studies addressing periprocedural pain.

Thus, the optimal anaesthetic procedure is still to be determined. Currently at our institution RF is performed as monitored sedation procedure using remifentanil infusion supplemented with midazolam boluses, when considered necessary. However, when using remifentanil and midazolam combination it is quite difficult to avoid too deep respiratory depression.

Dexmedetomidine is an α2-adrenoreceptor agonist with sedative, analgesic and anxiolytic effects, and it has more selective α2-adrenergic effect than clonidine. Dexmedetomidine has a great deal of potential in this arena given its analgesic and anxiolytic properties while preserving respiratory drive (Bergese SD et al., 2010).

All patients will receive dexmedetomidine 0.4 µg/kg/hr infusion from the start of procedure. The infusion will be continued during the whole RF procedure.

At the same time all patients will receive remifentanil infusion according to TCI (target controlled infusion) protocol. Plasma concentration target will be set from 0.5 ng/ml and, if necessary, will be increased to achieve a comfortable state of patient (Ramsey Sedation Scale: 2-3).

ELIGIBILITY:
Inclusion Criteria:

* liver or/and kidney cancer for which radiofrequency ablation procedure is planned
* signed informed consent form

Exclusion Criteria:

* patient refusal
* pregnancy
* known allergy to dexmedetomidine or remifentanil
* atrioventricular block grade II or III or other significant cardiac conduction disturbance
* stroke
* low blood pressure not responding to treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction With Sedation Technique | After completion of procedure (within 15 minutes)
  Rating of how satisfied the patient was with their sedation on a scale of 1-5 with 1 being very dissatisfied and 5 being extremely satisfied

SECONDARY OUTCOMES:
Vital signs: blood pressure, oxygen saturation, heart rate, breathing rate | During procedure and up to 2 hours stay at the post-anesthesia care unit
Ramsey Sedation Scale Score | During the procedure and up to 2 hours stay at the post-anesthesia care unit
  Rating of depth of sedation. Scale 1 - 6, 1 being wide awake and 6 being non-responsive
Maximal pain intensity | During procedure and up to 2 hours stay at the post-anesthesia care unit
  The 11-point Numerical Rating Scale (NRS) to assess periprocedural pain. Scale of 0-10, with 0:no pain and 10: pain as bad as it could be

CONTACTS AND LOCATIONS:
Overall Officials: Egidijus Semenas, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden; Mats Eriksson, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden